CLINICAL TRIAL: NCT00925574
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CNTO 1959 Following a Single Intravenous or a Single Subcutaneous Administration in Healthy Subjects and in Subjects With Moderate to Severe Psoriasis
Brief Title: A Study of the Safety and How the Body Affects a Drug (CNTO 1959) in Healthy Volunteers and in Patients With Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CR015817; CNTO1959PSO1001; CR015817
Record Dates: First submitted 2009-06-16; First posted 2009-06-22 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Psoriasis
Keywords: CNTO 1959; Healthy Volunteers; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: CNTO 1959; Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and how the body affects a drug (CNTO 1959) in healthy volunteers and in patients with psoriasis.

DETAILED DESCRIPTION:
CNTO 1959 is an experimental drug. In this study, CNTO 1959 will be tested to see if it may be useful in treating psoriasis. This disease causes inflammation of skin and nails. This is a Randomized (study drug assigned by chance), Double-blind (neither physician nor patient knows the name of the assigned drug), Placebo-controlled study of the experimental drug CNTO 1959 in both healthy patients as well as patients with psoriasis. This study will compare the effects (both good and bad) of CNTO 1959 to those of placebo. The purpose of this study is to evaluate the safety and potential side effects of CNTO 1959 given to healthy volunteers and patients with moderate to severe psoriasis. In addition, the investigators will measure how much study drug is in the blood following a dose of CNTO 1959, and determine if the body makes antibodies to it. (An antibody is a protein made by the body in response to a foreign substance). Safety assessments will be performed throughout the study and include obtaining and evaluating laboratory tests, vital signs (e.g., blood pressure), and the occurrence and severity of adverse events. This is the first time that CNTO 1959 will be studied in humans. There will be 2 parts to this study. The first part of this study will involve healthy volunteers, and the second part of the study will involve patients with psoriasis. About 47 healthy volunteers and 24 patients with moderate to severe psoriasis will take part in the study. Enrollment for the healthy volunteer part is closed as of 23SEP09. CNTO 1959 will be administered as either an intravenous (IV) infusion or subcutaneous (SC) injection. Duration of participation may be up to 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female with no clinically significant abnormalities and have a body weight of 50 to 100 kg (Enrollment of healthy volunteers closed on 23SEP09)
* Patients with moderate to severe psoriasis and have a body weight not greater than 120 kg.

Exclusion Criteria:

* Current or a history of any clinically significant medical illness or medical disorders the investigator considers should exclude the patient, including (but not limited to) cardiovascular disease, neuromuscular, hematological disease, respiratory disease, hepatic or GI disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* Known or recent history of alcohol or drug abuse
* Major or traumatic surgery within 12 weeks of screening
* Donated blood greater than 500 ml within 56 days of screening
* Pregnant or nursing
* Have recently received phototherapy or any systemic medications/treatments that could affect psoriasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-06-04 (Actual); Primary Completion 2010-10-11 (Actual); Study Completion 2010-10-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CNTO 1959 in healthy volunteers and patients with psoriasis. | Assessments will occur at each study visit and up to 24 weeks following administration of study agent

SECONDARY OUTCOMES:
Pharmacokinetics. | Assessments will occur at study visits through 24 weeks following administration of study agent.
Pharmacodynamics | Assessments will occur at study visits through 24 weeks following administration of study agent.
Immune Response | Assessments will occur at study visits through 24 weeks following administration of study agent.
Clinical Response | Assessments will occur at study visits through 24 weeks following administration of study agent.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (8):
- United States (8):
  - Los Angeles, California
  - San Diego, California
  - Miramar, Florida
  - Overland Park, Kansas
  - Baltimore, Maryland
  - St Louis, Missouri
  - New York, New York
  - Portland, Oregon

REFERENCES:
- See also: Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CNTO 1959 following a Single Intravenous or a Single Subcutaneous Administration in Healthy Subjects and in Subjects with Moderate to Severe Psoriasis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=193&filename=CR015817_CSR.pdf